CLINICAL TRIAL: NCT01672177
Title: Self Care for Older Persons in Singapore: An Intervention Study
Acronym: SCOPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Responsible Party: Principal Investigator, Dr. David Matchar, Professor and Director, Program in Health Services and Systems Research, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: MOE2010-T2-2-107
Record Dates: First submitted 2012-08-08; First posted 2012-08-24 (Estimated); Last update posted 2015-04-16 (Estimated); Status verified 2015-04

CONDITIONS: Health Services, Geriatric
Keywords: Geriatrics; Aged; Aging; Chronic disease; Self management
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Individuals in the control group will not receive any training.
- Intervention (Experimental): Individuals in the intervention group will receive two hour long weekly training sessions for seven to eight months. The content of the training focuses on health promotion, health seeking behaviours and chronic disease management.
  Interventions: Behavioral: Chronic disease self-management training

INTERVENTIONS:
Behavioral: Chronic disease self-management training — Those in the intervention group will receive two hour long weekly training sessions for seven-eight months (a total of 56 hours of training).
  Arms: Intervention

SUMMARY:
The main aim of the project is to evaluate a self-care intervention program aimed at enhancing the ability of mildly disabled and healthy older persons in Singapore to manage their health.

A secondary aim of the study is to evaluate the effectiveness of training community health workers located within Senior Activity Centres in Singapore to support the self-care capacity development amongst older persons in the locale.

DETAILED DESCRIPTION:
Singapore is facing a rapidly ageing population due to its changing demographics. One of the biggest challenges associated with older adults is providing them with adequate and sustainable health care. There are four main barriers that make it challenging to do so in this segment of the population: (1) Lack of knowledge of simple coping mechanisms and self care; (2) inadequate access to care and healthcare; (3) social, economic, and political exclusion; and (4) declining family support and strains on state services.

This proposal, is to conduct a randomized controlled trial that tests the impact of a state-of-the-art self care training program focused on teaching older adults how to manage their health and if present, their diabetes, hypertension or chronic obstructive pulmonary disease. The training focuses on health promotion, disease prevention, health seeking behavior, chronic disease management and empowerment. The study period is 18 months with measurements taken at baseline, 8 months and 18 months. Major events (stroke, myocardial infarction, end-stage renal disease, hospitalization, deaths) during the study will also be recorded. A questionnaire assessing functional status (IADL), quality of life (EQ5D), knowledge and attitude about health care, health seeking behavior, and health status (CIRS-G) will be used. Anthropometric measures will also be taken to better understand certain aspects related to the health and physical status of the participants as well as biomarkers such as the levels of glycosylated hemoglobin (HbA1c), cholesterol (total HDL), triglycerides, blood pressure and peak expiratory flow.

The main goal of the study is to improve each individual score and to measure improvement in overall quality of life and mental well-being. The total sample size for this pilot study is 400 older persons (above 55 years of age) randomly sampled from Tiong Bahru/Bukit Merah and Ang Mo Kio. The health care training will be based in Senior Activity Centres (SACs) located in HDB blocks. The investigators will select 12 SACs and randomly assign 6 SACs to the intervention group and 6 SACs to the control group. All twelve groups will receive a baseline assessment of physical and mental health status and a follow-up at 8 and 18 months. Two community health trainers (CHT) will be assigned to each of the intervention groups. These CHTs will have been trained by personnel at the Tsao Foundation to conduct the training protocol and collect data from participants. The intervention group will then receive the health care training once a week for 2 hours over a period of seven-eight months (56 hours total). The content of training materials focuses on health promotion, disease prevention, health seeking behavior, chronic disease management, and anti-stigmatization. In addition, each participant, regardless of randomization, will be given an event diary at baseline. The diary will be used to record any health related events that occur during the course of the study. Such events would include visits to GPs or traditional medicine practitioners, purchasing medications, hospitalization, etc.

The investigators hypothesize that the study will demonstrate the following: 1) Improve chronic disease outcomes for individuals presenting with these diseases: hypertension (20% decrease in systolic blood pressure), diabetes (1% decrease in HBA1C levels), and COPD (10% increase in peak expiratory flow) over the 18-month study period. 2) Improve quality of life of participants and their caregivers. 3) Improve knowledge, behaviours and attitudes towards health care utilization. 4) Develop a community health worker capacity in low-income settings. 5) Reduce the number of hospitalizations, outpatient and emergency visits in the intervention group.

This pilot study will also allow the investigators to test their methods for recruitment, training, and evaluation of the self-care training program. If successful, this study will provide evidence that older adults in the intervention group can more effectively manage their own health care and avert or delay the onset of disability compared to older adults in the control group. One of the long term goals is to replicate this study in Cambodia, India, Indonesia, and Vietnam. The investigators have identified academic and practice partners in each of these countries who have expressed an interest in the project and donors are awaiting the results from this pilot study before funding the regional components.

ELIGIBILITY:
Inclusion Criteria:

* Age 55 and above
* Age 21 or above for CHTs
* No cognitive impairment as justified by AMT
* No Activities of Daily Living (ADL)Limitations preventing them from coming to questionnaire interviews, health screenings, and/or weekly health trainings.
* Not severely ill ; not on dialysis, chemotherapy or psychiatric medication

Exclusion Criteria:

* Below 55 years of age
* Cognitively impaired
* Severely depressed
* With ADLs preventing them from coming to questionnaire interviews, health screenings, and/or weekly health trainings.
* Severely ill ; on dialysis, chemotherapy or psychiatric medication
* Those who refused to have their biomarkers taken (applies to both intervention and non-intervention group)

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2011-08; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Clinical Measures | 18 months
  The primary outcome measure is a composite of the change in the following measures: 1)Systolic BP; 2)HbA1C; and 3)normalized peak flow. The null hypothesis is that there is no difference between intervention and control in any of the measures.

SECONDARY OUTCOMES:
Improved Quality of Life | 18 months
  Improve quality of life of participants and their caregivers using a validated measure (EQ-5D).
Community Health Trainer | 18 months
  Develop a community health trainer capacity in low-income settings as assessed by numbers of individuals who successfully complete the health trainer education.
Healthcare Utilization | 18 months
  Reduce the number of hospitalizations, outpatient and emergency visits in the intervention group vs control.

CONTACTS AND LOCATIONS:
Overall Officials: David B Matchar, MD, Principal Investigator — Duke-NUS Graduate Medical School
Locations (12):
- Singapore (12):
  - Redhill SilverACE, Singapore
  - Moral Seniors Activity Centre (Redhill), Singapore
  - Moral Neighbourhood Link Bukit Merah View/Tanjong Pagar FSC, Singapore
  - Kreta Ayer Seniors Activity Centre (Chin Swee), Singapore
  - Sarah Seniors Activity Centre, Singapore
  - Kreta Ayer Senior Activity Centre (Jalan Kukoh), Singapore
  - AWWA Seniors Activity Centre, Singapore
  - Ang Mo Kio Family Services Centre, Singapore
  - Community Care Network Senior Activity Centre @Teck Ghee 420, Singapore
  - Care Corner Toa Payoh, Singapore
  - Lion Befrienders/TOUCH, Singapore
  - Moral Neighbourhood Link Telok Blangah, Singapore

REFERENCES:
- [Derived] Ng TKS, Wee HN, Ching J, Kovalik JP, Chan AW, Matchar DB. Plasma Acylcarnitines as Metabolic Signatures of Declining Health-Related Quality of Life Measure in Community-Dwelling Older Adults: A Combined Cross-sectional and Longitudinal Pilot Study. J Gerontol A Biol Sci Med Sci. 2024 Mar 1;79(3):glac114. doi: 10.1093/gerona/glac114. PMID 35605263
- [Derived] Ng TKS, Matchar DB, Sultana R, Chan A. Effects of Self-Care for Older PErsons (SCOPE) on Functional and Physiological Measures: A Cluster Randomized Controlled Trial. J Clin Med. 2020 Mar 24;9(3):885. doi: 10.3390/jcm9030885. PMID 32213860
- [Derived] Chan A, Matchar DB, Tsao MA, Harding S, Chiu CT, Tay B, Raman P, Pietryla Z, Klein MK, Haldane VE. Self-Care for Older People (SCOPE): a cluster randomized controlled trial of self-care training and health outcomes in low-income elderly in Singapore. Contemp Clin Trials. 2015 Mar;41:313-24. doi: 10.1016/j.cct.2015.01.001. Epub 2015 Jan 10. PMID 25583272